CLINICAL TRIAL: NCT06303479
Title: The Effect of Telerehabilitation-Based Breathing Exercise Programs With and Without Instruments on Lung Capacity
Brief Title: The Effect of Telerehabilitation-Based Respiratory Exercise Programs on Lung Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Voldyne_Tele
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-12

CONDITIONS: Breathing Exercises; Telerehabilitation
Keywords: spirometry; physical activity; lung volume
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrumental breathing exercise group (Experimental): Instrumental breathing exercise group consisting of 13 healthy adults between the ages of 18-30
  Interventions: Other: Instrumental breathing exercise group
- Non-Instrumental breathing exercise group (Experimental): Non-Instrumental breathing exercise group consisting of 13 healthy adults between the ages of 18-30
  Interventions: Other: Non-Instrumental breathing exercise group

INTERVENTIONS:
Other: Non-Instrumental breathing exercise group — Before starting the exercises, participants will be told about diaphragmatic breathing exercises, maximum inspiratory holding technique and thoracic expansion exercises through the Zoom program by telerehabilitation method, and people will be checked by the physiotherapist who manages the program during the practice. The program will last for 8 weeks and will be planned to be implemented 5 days a week in total, including 2 days of telerehabilitation, 3 days of home program. The participant will be asked to start the exercises in a reclining position with his back to the chair. He will be asked to place his right hand on his upper abdomen and his left hand on the upper side of his chest. In each session, the exercises will be performed with 1 set of 10 repetitions for each of the diaphragmatic breathing and thoracic expansion exercises and will progress with progression.
  Arms: Non-Instrumental breathing exercise group
Other: Instrumental breathing exercise group — The volume-oriented spirometer works with pressure and its indicator changes during breathing. When the participants breathe, the pressure in the tube decreases and the piston of the spirometer rises. The inhaled breath volume is seen at the top of the piston. In our study, participants will be told about the exercises through the Zoom program using the telerehabilitation method, and people will be checked by the responsible physiotherapist who manages the program during the application. The program will last for 8 weeks, 2 days of telerehabilitation, 3 days of home program will be planned to be implemented 5 days a week in total. Participants will be instructed to breathe up to their total lung capacity and maintain continuous inspiration for at least 3 seconds. The exercises will start with 1 set of 15 repetitions and the program will progress with progression.
  Arms: Instrumental breathing exercise group

SUMMARY:
It is a prospective randomized controlled trial. In this project, it is aimed to examine the effect of telerehabilitation-based instrumental and noninstrumental respiratory exercise program on lung capacities. For this reason;

* Contributing to the literature by comparing the effect of breathing exercises with and without instruments on lung capacities,
* It is aimed to be a resource for the effective use of respiratory exercise, which has a high effect on lung capacities, in treatment.

In addition, with the data obtained, it is aimed to decide and apply the exercise that is more effective in the treatment of respiratory diseases quickly.

Socio-demographic data will be questioned by using the Demographic Data Form; participants, age, gender, height, weight, marital status, smoking and alcohol use, presence of disease, whether they are included in a different exercise program, dyspnea, severe nausea and vomiting. The cases will be randomized into two groups: non-instrumented breathing exercises group and instrumented breathing exercises group. The physical activity status of the individuals participating in the study will be questioned using the International Physical Activity Questionnaire-Short Form (IPAQ-SF) at the beginning and end of the study. Pulmonary Function Test (PFT) will be used to measure the lung capacity of the participants.

Instrumented breathing exercises will be performed for 8 weeks, 2 days a week with the telerehabilitation program, 3 days a week as a home program, 5 days a week in total, starting with 1 set of 15 repetitions and the program will progress with progression. Diaphragmatic breathing and thoracic extension exercises will be applied as non-instrumented breathing exercises. For 8 weeks, 2 days a week with telerehabilitation method, 3 days a week as a home program, 5 days a week in total, 1 set of 10 repetitions for each exercise and the program will progress with progression. At the end of 8 weeks, all evaluations of the participants in both groups will be repeated.

DETAILED DESCRIPTION:
Breathing exercises are one of the components of pulmonary rehabilitation that have been widely used in clinical practice for many years. Exercises such as pursed lip breathing, local expansion, diagraphmatic breathing, holding at maximum inspiration are some of the breathing exercises in the literature. Such breathing exercises dilate the airways, facilitate gas exchange in the alveoli, increase the amount of oxygen reaching the cells, and normalize respiratory functions. Diaphragmatic breathing is a technique that uses the contraction of the diaphragm muscle to increase the length of the diaphragm and the efficiency of breathing, resulting in more efficient expiration. Studies have shown that diaphragmatic breathing reduces respiratory workload and dyspnea, increases respiratory efficiency and exercise tolerance, and improves minute ventilation by reducing the number of breaths. The aim of respiratory exercises is to maintain and improve respiratory function and to increase the amount of air entering and leaving the lungs. The amount of incoming and outgoing air is called lung volume and capacity. Lung volumes and capacities; forced expiratory volume in one second (FEV1), forced vital capacity (FVC), Tiffeneau index (FEV1\FVC), peak expiratory flow (PEF) will be compared.

There are also many therapeutic devices developed among respiratory exercises. The incentive spirometer is one of these exercise devices. The incentive spirometer can be used for two different purposes: volume-oriented or flow-oriented. Studies have shown that volume-oriented devices are more effective in improving respiratory parameters than flow-oriented devices. In the literature, it is stated that the use of spirometers increases lung capacities, provides more comfortable air entry into the alveoli and facilitates gas exchange.

Telerehabilitation method is defined as the remote delivery of rehabilitation services by rehabilitation specialists with certain procedures and protocols using tools such as information and communication technologies. With telerehabilitation, it is aimed to follow patients at home, to carry rehabilitation services far away and to provide health services directly where the patient is.

In this project, it is aimed to examine the effect of telerehabilitation-based instrumental and noninstrumental respiratory exercise program on lung capacities. In the literature, there is no study comparing the efficacy of telerehabilitation-based instrumental and noninstrumental respiratory exercise program on healthy young adults. Thus, this project will contribute to the literature and will be a preliminary study for advanced research in this field.

ELIGIBILITY:
Inclusion Criteria:

* Female/male young adult between the ages of 18-30 December,
* Who volunteered to participate in the study,
* Without a known disease
* Volunteers who do not have psychological, cognitive and emotional problems

Exclusion Criteria:

* Cigarette and alcohol users
* People with severe cardiopulmonary disorders
* People with postural disorders (such as scoliosis,kyphosis...)
* Unstable angina, has it been recently, pulmonary embolism
* People with obesity/diabetes
* Mental or cognitive impairment that will affect mental cooperation
* People with severe nausea, vomiting attacks
* People with dyspnea
* People with orthopedic disorders that will affect exercise performance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-09-29 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test for FEV1 | At baseline and 8 weeks
  Pulmonary function test will be performed with desktop type spirometry. The FEV1 value will be calculated.
Pulmonary Function Test for PEF | At baseline and 8 weeks
  Pulmonary function test will be performed with desktop type spirometry. The PEF value will be calculated.
Pulmonary Function Test for FEV1/FVC | At baseline and 8 weeks
  Pulmonary function test will be performed with desktop type spirometry. The FEV1/FVC value will be calculated.
Pulmonary Function Test for FVC | At baseline and 8 weeks
  Pulmonary function test will be performed with desktop type spirometry. The FVC value will be calculated.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | At baseline and 8 weeks
  IPAQ-SF is a form designed to measure physical activity among individuals. It includes leisure time physical activities, home and garden activities, work-related physical activities, transportation-related physical activities. Physical activity status will be determined by this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nur AYYILDIZ, Student, Study Chair — Saglik Bilimleri Universitesi; Beyzanur YEŞİLYURT, Student, Study Chair — Saglik Bilimleri Universitesi; Fulya KARAAHMETOĞLU, PhD (c), Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)